CLINICAL TRIAL: NCT05042089
Title: Predictive Features of Pre-operative Computed Tomography and Magnetic Resonance Imaging for Advanced Disease in Renal Cell Carcinoma
Brief Title: Predictive Imaging Features in Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, selman unal, Principal Investigator, Ankara Yildirim Beyazıt University
Other Study IDs: AnkaraYBU-URO-SU-03
Record Dates: First submitted 2021-09-04; First posted 2021-09-13 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Renal Malignant Tumor
Keywords: Renal Cell Carcinoma; Tomography; Magnetic resonance imaging
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pathological tumor stage 1-2 (pT1-2): Stage pT1 and pT2 according to pathology results of patients who underwent partial or radical nephrectomy.
  Interventions: Other: No intervention will be applied.
- pathological tumor stage ≥pT3a: Stage ≥pT3a according to pathology results of patients who underwent partial or radical nephrectomy.
  Interventions: Other: No intervention will be applied.

INTERVENTIONS:
Other: No intervention will be applied. — The preoperative imaging of the participants, who were grouped according to the postoperative pathology results, will be examined.

SUMMARY:
The investigators aimed to evaluate the role of some findings that can be detected in preoperative radiological imaging of kidney masses in predicting locally advanced disease.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) is one of the most common urinary system cancers and accounts for 3% of all cancers. With the frequent use of imaging methods most renal masses are detected localized. The standard treatment option in localized RCC is radical nephrectomy (RN) or nephron-sparing surgery (NSS). NSS is preferred when appropriate in patients with tumor stage 1 (T1) and has been shown to be comparable to RN in terms of oncologic outcomes. Although there is no prospective randomized study comparing NSS with RN in terms of oncological and renal functions in T2 patients, there are retrospective studies conducted to date. According to the current European urology guideline, the standard approach in patients with T2 and above is RN. Pre-operative clinical staging is performed with computed tomography (CT) or magnetic resonance imaging (MRI), and patients may develop local recurrence despite surgical procedures based on clinical stage. Pre-operative the patient and in the management of local disease. In clinical practice, pre-operative CT and MRI provide information about tumor size, tumor localization, presence of tumor invasion into vascular structures and adjacent organs. However, apart from these frequently reported findings, there are CT and MRI findings that can be used to predict advanced disease. In the 2017 Tumor, node, metastasis (TNM) classification, invasion of the pelvicalyceal system, perirenal or renal sinus fat invasion has been included in the T3a category. There are studies evaluating predictive value of CT to indicate renal sinus fat or perirenal fat invasion. Although not in the standard TNM classification, it has been shown that renal capsule invasion is an independent prognostic variable for advanced disease and can be detected on CT. On the other hand, it has been indicated that thickening of the Gerota's fascia, the presence of enlarged collateral vessels, and the presence of intra-tumoral necrosis may be imaging findings that can be used to predict advanced disease. The investigators think that the markers evaluated so far in pre-operative imaging and some additional markers may predict advanced disease in RCC. The investigators also think that the predictive value of MRI may be higher than CT. Therefore, in this study the investigators evaluated some predictive features (Renal capsule invasion, perirenal fat invasion, thickening of the Gerota's fascia, presence of enlarged collateral vessels, tumor necrosis, perinephric stranding) of pre-operative computed tomography and magnetic resonance imaging for advanced disease in renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* patients operated for kidney mass
* patients with preoperative CT or MRI imaging

Exclusion Criteria:

* metastatic RCC
* who had undergone surgery on the same side before kidney mass due to other urological pathologies
* who had pathology results other than RCC (oncocytoma, etc.)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 20-80 years who have a renal mass detected by CT or MR imaging in the urology outpatient clinic and undergo partial or radical nephrectomy.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Renal capsule invasion | 1 month
  Whether there was a difference between the two groups in terms of the presence of pre-operative imaging (CT and MRI) renal capsule invasion.
Perirenal fat tissue invasion | 1 month
  Whether there was a difference between the two groups in terms of the presence of pre-operative imaging (CT and MRI) perirenal fat tissue invasion
Thickening of the Gerota's fascia | 1 month
  Whether there was a difference between the two groups in terms of the presence of pre-operative imaging (CT and MRI) thickening of the Gerota's fascia.

CONTACTS AND LOCATIONS:
Overall Officials: Selman Unal, Principal Investigator — Ankara Yildirim Beyazit University School of Medicine, Department of Urology
Locations (1):
- Ankara Yildirim Beyazit University, Schhol of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No